CLINICAL TRIAL: NCT06782516
Title: Native-RISE (Risk Identification for Suicide and Enhanced Care)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00026145
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Native-RISE Model is a predictive algorithm for suicide risk in Native American populations. The algorithm was developed based on analysis of over 330,000 visits and designed to identify people at risk of a suicide attempt or death within 90 days of the last visit. The evaluation of the model initial results have been published with the model having an area under the ROC (AUROC) 0.83 [0.80-0.86]) and performing better than existing care (AUROC 0.64 [0.61-0.67]).
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Case Managers WITH algorithm AND with provider risk notification (SI/SA/Binge/NSSI) (Experimental): Case Managers who see the algorithm classification + IHS provider risk notification & resource card distribution. These participants present with suicide ideation (SI), suicide attempt (SA), binge substance use (Binge), or non-suicidal self injury (NSSI).
  Interventions: Device: System of Care - combination of algorithm and Brief Contact Intervention
- Case Managers withOUT algorithm AND with provider risk notification (SI/SA/Binge/NSSI) (Active Comparator): Case Managers who do NOT see the algorithm classification + IHS provider risk notification & resource card distribution. These participants present with suicide ideation (SI), suicide attempt (SA), binge substance use (Binge), or non-suicidal self injury (NSSI).
  Interventions: Behavioral: Active Comparator - Provider notification of risk status
- Case Managers WITH algorithm AND provider risk notification (high risk history, no SI/SA/Binge/NSSI (Experimental): Case Managers who see the algorithm classification + provider risk notification; participants get resource card distribution. High risk participants based on algorithm classification.
  Interventions: Device: System of Care - combination of algorithm and Brief Contact Intervention
- Provider risk notification alone (high risk history, without SI/SA/Binge/NSSI) (Active Comparator): Provider risk notification alone; participants get resource card distribution. High risk participants based on algorithm classification.
  Interventions: Behavioral: Active Comparator - Provider notification of risk status

INTERVENTIONS:
Device: System of Care - combination of algorithm and Brief Contact Intervention — Case managers see the Native-RISE algorithm classification and Clinical Providers receive a risk notification. A resource card is provided to the participant.
  Arms: Case Managers WITH algorithm AND provider risk notification (high risk history, no SI/SA/Binge/NSSI; Case Managers WITH algorithm AND with provider risk notification (SI/SA/Binge/NSSI)
Behavioral: Active Comparator - Provider notification of risk status — Clinical Providers receive a risk notification and a resource card is provided to the participant.
  Arms: Case Managers withOUT algorithm AND with provider risk notification (SI/SA/Binge/NSSI); Provider risk notification alone (high risk history, without SI/SA/Binge/NSSI)

SUMMARY:
The goal of this research is to test a systems-level suicide prevention strategy, Native-RISE (Risk Identification for Suicide and Enhanced care), that combines predictive analytics and brief contact interventions (BCIs) to reduce suicide in health systems serving Native Americans (NAs). This project aims to prove the effectiveness and scalability of Native-RISE within three Indian Health Service (IHS) health care clinics (Whiteriver, Chinle and Shiprock) already implementing suicide prevention programs and serving the White Mountain Apache Tribe (WMAT) and Navajo Nation (NN).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75
* Visit at least one of the three participating IHS clinics
* Identified as at risk of suicide by either an existing method or the new Native-RISE risk model algorithm

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1687 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of suicide attempts among individuals flagged at elevated risk | 12 months
  Rate of suicide attempts among individuals flagged at elevated risk is tracked through International Classification of Diseases (ICD) codes and chief complaints as recorded in the participating health system.

SECONDARY OUTCOMES:
Number of contacts with Case Managers (Reach of Brief Contact Interventions (BCI)) | 12 months
  Reach of BCI is defined as at least three or more contacts with Case Managers within the first year following identification of elevated risk.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Haroz, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Chinle Navajo Nation Center for Indigenous Health, Chinle, Arizona
  - Whiteriver Center for Indigenous Health, Whiteriver, Arizona
  - Shiprock Center for Indigenous Health, Shiprock, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haroz EE, Rebman P, Goklish N, Garcia M, Suttle R, Maggio D, Clattenburg E, Mega J, Adams R. Performance of Machine Learning Suicide Risk Models in an American Indian Population. JAMA Netw Open. 2024 Oct 1;7(10):e2439269. doi: 10.1001/jamanetworkopen.2024.39269. PMID 39401036
- [Background] Adams R, Haroz EE, Rebman P, Suttle R, Grosvenor L, Bajaj M, Dayal RR, Maggio D, Kettering CL, Goklish N. Developing a suicide risk model for use in the Indian Health Service. Npj Ment Health Res. 2024 Oct 16;3(1):47. doi: 10.1038/s44184-024-00088-5. PMID 39414996